CLINICAL TRIAL: NCT05645666
Title: The Effectiveness of Well-being Therapy on Mental Health and Self-efficacy of Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Isfahan (Khorasgan) Branch (Other)
Responsible Party: Principal Investigator, Arezoo Ziaei, M.A Student, Islamic Azad University, Isfahan (Khorasgan) Branch
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13115
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well being therapy (Experimental): The group of 16 which recieved well-being therapy
  Interventions: Behavioral: Well-being therapy
- Control group (No Intervention): The group of 16 which did not recieve well-being therapy

INTERVENTIONS:
Behavioral: Well-being therapy — Well-being therapy is a short-term, organized and problem-oriented treatment program that is based on Riff's psychological well-being model. Its purpose is to help patient in order to improve His/her functions in six dimensions; personal growth, environmental mastery, purposefulness of life, and autonomy, self-acceptance and positive relationships with others Therapists help patients find well-being experiences in their present and past lives and pay attention to these experiences, no matter how small or short they are.
  Arms: Well being therapy

SUMMARY:
Ulcerative colitis (UC) is a chronic and lifelong disease that causes disabilities for sufferers and causes mental health disorders in the patients. For this reason, it is important to know which psychotherapy is more effective for UC patient's problems, and since no research has been done on the effectiveness of well-being therapy on the mental health problems of these patients, this research can help psychologists and other specialists in this field to help patients with UC and other chronic disease.

The present study is conducted with the aim of determining the effectiveness of mental well-being on the mental health and quality of life of patients with ulcerative colitis. The research method was a semi-experimental type with a pre-test-post-test design with a control group. The study population included all patients with ulcerative colitis who were previously diagnosed with ulcerative colitis by a gastroenterologist and referred to one of the gastroenterology centers for treatment. The criteria for entering the patients into the study were: definitive diagnosis of ulcerative colitis according to the opinion of a gastroenterologist, consent to participate in the study, having at least a high-school education and an age range of 18 to 60 years. The patients who were excluded from the study were: patients who have acute Psychiatric or other medical disorders , patients who have participated in counseling or psychotherapy sessions in the last six months and patients who lose motivation to participate in the interview or are absent for more than two sessions. The convenience sampling method was used. The list of patients with inflammatory bowel diseases was provided to the researcher after the consent of the head of the Digestive Disease Research Institute. 300 ulcerative colitis patients of this list were contacted according to the criteria for entering the study, and they were invited to participate in the treatment sessions after a brief explanation about the objectives of the sessions, sessions duration and time. Finally, 32 patients volunteered and were randomly assigned to one of the following groups:

16 people (9 women and 7 men) were in the well-being therapy group and 16 people (8 men and 8 women) were in the control group. In the post-test phase, one person in the study group stopped working, and in the follow-up phase, which was done 6 months later , the study did face any shortages.

ELIGIBILITY:
Inclusion Criteria:

- definitive diagnosis of ulcerative colitis according to the opinion of a gastroenterologist, consent to participate in the study, having at least a high-school education and an age range of 16 to 60 years.

Exclusion Criteria:

patients who have acute Psychiatric or other medical disorders , patients who have participated in counseling or psychotherapy sessions in the last six months and patients who lose motivation to participate in the interview or are absent for more than two sessions

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Pre-test level | Immediately after the intervention
  The results demonstrated that the effectiveness of this treatment on the level of self-efficacy and mental health was significant in the pretest phase.
Follow-up level | 6 months after the intervention
  The results demonstrated that the effectiveness of this treatment on the level of self-efficacy and mental health was significant in the follow-up phase

CONTACTS AND LOCATIONS:
Overall Officials: Ziaei, Principal Investigator — M.A student, Department of Educational Science and Psychology, Isfahan(Khorasgan) Branch, Islamic Azad University
Locations (1):
- Educational Science and Psychology, Isfahan, Iran

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391